CLINICAL TRIAL: NCT05537493
Title: Efficiency of Telerehabilitation in Patients Operated With the Diagnosis of Distal Radius Fracture
Brief Title: Tele-rehabilitation in Patients Operated for Distal Radius Fracture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahi Evran University Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Levent Horoz, Assist Prof, Ahi Evran University Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KAEK_2022-09/96
Record Dates: First submitted 2022-09-09; First posted 2022-09-13 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Distal Radius Fracture
Keywords: telerehabilitation; distal radius fracture; functionality
MeSH Terms: conditions — Wrist Fractures | interventions — Telerehabilitation

STUDY DESIGN:
Intervention Model Description: Romdomised controlled
Who Masked: Outcomes Assessor
Masking Description: Evaluator is blind to study groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitation (Experimental): Videos of the exercises they will do via whatsapp will be sent to the telerehabilitation group. Again, in telerehabilitation, whatapp application will be made in the form of videoconference. Rehabilitation program will be applied to the patients 4 times a week for 6 weeks.
  Interventions: Other: Telerehabilitation
- Face to face (Active Comparator): A rehabilitation program will be applied to the Face to Face rehabilitation group by a physiotherapist in the hospital for a total of 30 sessions per week for 6 weeks.
  Interventions: Other: Face to face

INTERVENTIONS:
Other: Telerehabilitation — It will be followed by exercising on whatsapp
  Arms: Telerehabilitation
Other: Face to face — It will be followed by face to face
  Arms: Face to face

SUMMARY:
It was designed as a randomized controlled prospective. After 2 weeks of splint follow-up, the splints of the patients who were operated due to distal radius fracture and volar plate were applied will be removed and included in the physical therapy program. The measurements and scores of the patients at the time of removal of the splint will be recorded. Patients' non-injured contralateral extremity data will also be recorded. The dominant party will be registered. Preoperative fracture classification of the patients, reduction parameters after surgery, waiting time for post-fracture surgery, pre-fracture chronic diseases, cognitive disorders, psychiatric disease histories, whether the patients lived alone at home or not will be recorded. Patients will be randomized with the help of a free computer aided numerator. The patients will be divided into two groups and conventional face-to-face rehabilitation will be applied to one group, and the previously planned tele-rehabilitation program will be applied to the other group.

DETAILED DESCRIPTION:
It was designed as a randomized controlled prospective. After 2 weeks of splint follow-up, the splints of the patients who were operated due to distal radius fracture and volar plate were applied will be removed and included in the physical therapy program. The measurements and scores of the patients at the time of removal of the splint will be recorded. Patients' non-injured contralateral extremity data will also be recorded. The dominant party will be registered. Preoperative fracture classification of the patients, reduction parameters after surgery, waiting time for post-fracture surgery, pre-fracture chronic diseases, cognitive disorders, psychiatric disease histories, whether the patients lived alone at home or not will be recorded. Patients will be randomized with the help of a free computer aided numerator. The patients will be divided into two groups and conventional face-to-face rehabilitation will be applied to one group, and the previously planned tele-rehabilitation program will be applied to the other group. Videos of the exercises they will do via whatsapp will be sent to the telerehabilitation group. Again, in telerehabilitation, whatapp application will be made in the form of videoconference. Rehabilitation program will be applied to the patients 4 times a week for 6 weeks. Rehabilitation will be applied to the groups by the same person. At the end of the rehabilitation program, the first measurements of the patients will be taken. The third measurement of the patients will be taken at the 3rd month after the surgery. Among the parameters to be checked, grip strength, wrist range of motion, Shortened Disabilities of the Arm, Shoulder, and Hand (QuickDASH) and Patient-Rated Wrist Evaluation (PRWE) questionnaire, VAS scale will be used. Solid side values will be recorded. Tele-rehabilitation satisfaction survey will be applied in the 3rd month controls of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Application of volar plate for distal radius fracture
* Patients not having undergone any surgery on that extremity before, not having an extremity defect that prevents rehabilitation
* Patients with normal pre-fracture cognitive functions
* Patients without major postoperative complications

Exclusion Criteria:

* Polytrauma
* Previous extremity-related surgery
* Injury in more than one anatomical region in the relevant extremity
* Patients living alone at home
* Malignancy, presence of known rheumatological disease, pregnancy
* Patients receiving any treatment other than the planned treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2022-05-25 (Actual); Primary Completion 2023-04-11 (Actual); Study Completion 2023-05-11 (Actual)

PRIMARY OUTCOMES:
Wrist joint range of motion | 0 day
  Wrist joint range of motion (ROM) measurement with goniometer is the most commonly used method that provides objective evaluation and error-free measurement in clinical practice. In our study, wrist ROM measurements will be made with a goniometer using the neutral zero method. This method is a painless and non-invasive measurement method.
Wrist joint range of motion | 6 th week
  Wrist joint range of motion (ROM) measurement with goniometer is the most commonly used method that provides objective evaluation and error-free measurement in clinical practice. In our study, wrist ROM measurements will be made with a goniometer using the neutral zero method. This method is a painless and non-invasive measurement method.
Wrist joint range of motion | 12 th week
  Wrist joint range of motion (ROM) measurement with goniometer is the most commonly used method that provides objective evaluation and error-free measurement in clinical practice. In our study, wrist ROM measurements will be made with a goniometer using the neutral zero method. This method is a painless and non-invasive measurement method.Likert scale. Patients are asked to indicate the level of pain, with 0 points as no pain, 5 points as moderate pain, and 10 points as unbearable pain. Increased scores indicate higher pain level.
Environmental Measurement | 0 day
  Environmental Measurement; Both hands and wrists of the patient will be measured with the figure of eight method with the help of a tape measure. The cm difference between both upper extremities will be recorded.
Environmental Measurement | 6 th week
  Environmental Measurement; Both hands and wrists of the patient will be measured with the figure of eight method with the help of a tape measure. The cm difference between both upper extremities will be recorded.
Environmental Measurement | 12th week
  Environmental Measurement; Both hands and wrists of the patient will be measured with the figure of eight method with the help of a tape measure. The cm difference between both upper extremities will be recorded.
Quick-DASH | 0 day
  The short version of the Arm, Shoulder and Hand Questionnaire (Quick-DASH) Disability will be used to evaluate the functional status of patients. Quick-DASH is a self-report questionnaire designed to measure physical function and symptoms in people with upper extremity musculoskeletal conditions. Turkish validity reliability was done
Quick-DASH | 6th week
  The short version of the Arm, Shoulder and Hand Questionnaire (Quick-DASH) Disability will be used to evaluate the functional status of patients. Quick-DASH is a self-report questionnaire designed to measure physical function and symptoms in people with upper extremity musculoskeletal conditions. Turkish validity reliability was done
Quick-DASH | 12th week
  The short version of the Arm, Shoulder and Hand Questionnaire (Quick-DASH) Disability will be used to evaluate the functional status of patients. Quick-DASH is a self-report questionnaire designed to measure physical function and symptoms in people with upper extremity musculoskeletal conditions. Turkish validity reliability was done
Coarse Grip Strength | 0 day
  Coarse Grip Strength: Coarse grip; It is caused by the combined activities of the intrinsic and extrinsic muscles of the hand. In our study, Jamar dynamometer was used for the evaluation of rough grip strength. The digital handheld dynamometer can measure in pounds and kg.
Coarse Grip Strength | 6th week
  Coarse Grip Strength: Coarse grip; It is caused by the combined activities of the intrinsic and extrinsic muscles of the hand. In our study, Jamar dynamometer was used for the evaluation of rough grip strength. The digital handheld dynamometer can measure in pounds and kg.
Coarse Grip Strength | 12th week
  Coarse Grip Strength: Coarse grip; It is caused by the combined activities of the intrinsic and extrinsic muscles of the hand. In our study, Jamar dynamometer was used for the evaluation of rough grip strength. The digital handheld dynamometer can measure in pounds and kg.
Patient-Rated Wrist Evaluation (PRWE) questionnaire | 0 day
  Patient-Rated Wrist Evaluation (PRWE) questionnaire: PRWE is a 15-item questionnaire designed to measure wrist pain and disability in activities of daily living. PRWE consists of 2 subscales that assess patients' wrist pain levels and disability. The PAIN subscale (0 = no pain, 10 = worst ever) and the FUNCTION subscale (0 = no difficulty, 10 = unable). Turkish validity and reliability was established.
Patient-Rated Wrist Evaluation (PRWE) questionnaire | 6th day
  Patient-Rated Wrist Evaluation (PRWE) questionnaire: PRWE is a 15-item questionnaire designed to measure wrist pain and disability in activities of daily living. PRWE consists of 2 subscales that assess patients' wrist pain levels and disability. The PAIN subscale (0 = no pain, 10 = worst ever) and the FUNCTION subscale (0 = no difficulty, 10 = unable). Turkish validity and reliability was established.
Patient-Rated Wrist Evaluation (PRWE) questionnaire | 12th week
  Patient-Rated Wrist Evaluation (PRWE) questionnaire: PRWE is a 15-item questionnaire designed to measure wrist pain and disability in activities of daily living. PRWE consists of 2 subscales that assess patients' wrist pain levels and disability. The PAIN subscale (0 = no pain, 10 = worst ever) and the FUNCTION subscale (0 = no difficulty, 10 = unable). Turkish validity and reliability was established.
pinch grip strength. | 0 day
  Pinchmeter device will be used to measure the pinch grip strength. The pinchmeter will be placed between the tip of the participant's thumb and the tip of the index finger to measure in the standard position recommended by the American Association of Hand Therapists (AETD).
pinch grip strength. | 6 th week
  Pinchmeter device will be used to measure the pinch grip strength. The pinchmeter will be placed between the tip of the participant's thumb and the tip of the index finger to measure in the standard position recommended by the American Association of Hand Therapists (AETD).
pinch grip strength. | 12th week
  Pinchmeter device will be used to measure the pinch grip strength. The pinchmeter will be placed between the tip of the participant's thumb and the tip of the index finger to measure in the standard position recommended by the American Association of Hand Therapists (AETD).

CONTACTS AND LOCATIONS:
Overall Officials: Levent Horoz, Asisst Prof, Principal Investigator — Kirsehir Ahi Evran Universitesi
Locations (1):
- Ahi Evran University, Kirşehir, City Centre, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bini SA, Mahajan J. Clinical outcomes of remote asynchronous telerehabilitation are equivalent to traditional therapy following total knee arthroplasty: A randomized control study. J Telemed Telecare. 2017 Feb;23(2):239-247. doi: 10.1177/1357633X16634518. Epub 2016 Jul 9. PMID 26940798
- [Background] Kane LT, Thakar O, Jamgochian G, Lazarus MD, Abboud JA, Namdari S, Horneff JG. The role of telehealth as a platform for postoperative visits following rotator cuff repair: a prospective, randomized controlled trial. J Shoulder Elbow Surg. 2020 Apr;29(4):775-783. doi: 10.1016/j.jse.2019.12.004. PMID 32197766
- [Background] Pastora-Bernal JM, Martin-Valero R, Baron-Lopez FJ, Moyano NG, Estebanez-Perez MJ. Telerehabilitation after arthroscopic subacromial decompression is effective and not inferior to standard practice: Preliminary results. J Telemed Telecare. 2018 Jul;24(6):428-433. doi: 10.1177/1357633X17706583. Epub 2017 Apr 27. PMID 28449618